CLINICAL TRIAL: NCT05140824
Title: A Multicenter, Randomized, Double-blind, Placebo-Controlled, Phase 1 Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of Single and Multiple Doses of TJ202 in Patients With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety, Tolerability, and PK Profile of Single and Multiple Doses TJ202 in Patient With Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company development strategy adjustment
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJ202001SLE101
Record Dates: First submitted 2021-11-04; First posted 2021-12-01 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Evaluate the Safety, Tolerability; A Multicenter, Randomized, Double-blind, Placebo-Controlled, Phase 1 Clinical Study
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 0.9% sodium chloride solution
  Interventions: Drug: Placebo
- TJ202 (Experimental): TJ202 injection
  Interventions: Biological: TJ202 injection

INTERVENTIONS:
Drug: Placebo — 0.9% sodium chloride solution
  Arms: Placebo
Biological: TJ202 injection — TJ202 injection
  Arms: TJ202

SUMMARY:
A Multicenter, Randomized, Double-blind, Placebo-Controlled, Phase 1 Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of Single and Multiple Doses of TJ202 in Patients with Systemic Lupus Erythematosus

ELIGIBILITY:
Inclusion Criteria (subjects must meet all the following criteria for inclusion in this study):

Single Dose:

1. Male or female, 18-65 years old (inclusive), weight of ≥ 45 kg.
2. Definite diagnosis of systemic lupus erythematosus (see Annex 3. SLE Classification Criteria by SLICC 2012 for diagnostic criteria), and an SLE disease activity index (SLEDAI) score of < 15 (see Annex 4. SLE Disease Activity Score [SLEDAI-2000] for scoring criteria) . A positive antinucleus antibody (ANA) test result.
3. If a subject is receiving SLE treatment, a stable SLE regimen must be maintained up to the date of the first dose of study drug (the permitted medications and their maximum doses are as follows):

   * Glucocorticoids: prednisone 10 mg/day or other glucocorticoids with an equivalent dose. It should be stable for at least 4 weeks prior to receiving the first dose of study drug.
   * Other immunosuppressive drugs alone or in combination with glucocorticoids include the following: azathioprine (maximum dose of 100 mg/day), methotrexate (maximum dose of 15 mg/week), mycophenolate mofetil (maximum dose of 1500 mg/day), tripterygium wilfordii polyglycosides (maximum dose of 60 mg/day), leflunomide (maximum dose of 20 mg/day), tacrolimus (maximum dose of 4 mg/day), ciclosporin (maximum dose of 100 mg/day). The above medications should be used for at least 12 weeks and stable for at least 4 weeks prior to receiving the first dose of study drug.
   * Hydroxychloroquine: The maximum allowable dose is 400 mg/day, and combination with the immunosuppressants listed above is allowed. It should be used for at least 12 weeks and the dose should be stable for at least 4 weeks prior to receiving the first dose of study drug.
4. The subject is willing to participate in the study and voluntarily sign the ICF.
5. Subjects of childbearing potential or subjects with a partner of childbearing potential must agree to use effective contraceptive measures throughout the study (except oral estrogens, estrogenic vaginal ring, etc., refer to Annex 5. Contraceptive Measures, Definitions of Women of Childbearing Potential and Contraception Requirements for optional contraceptive methods).

   Multiple Doses: in addition to the single-dose inclusion criteria, subjects should meet the following criteria
6. dsDNA antibody titer (ELISA) greater than or equal to 1.5 times the upper limit of normal (ULN).

Exclusion Criteria (subjects who meet any of the following criteria will be excluded from the study):

1. Central nervous system (CNS) diseases: active central nervous system lupus (including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident, encephalitis, or CNS vasculitis), visual disturbance, cranial neuropathy within 60 days prior to screening, with intervention required.
2. Renal disorders: nephrotic syndrome (protein urine > 3.5 g/24 h) within 30 days prior to screening, or requiring protocol-prohibited medications (such as intravenous cyclophosphamide) for active nephritis, or requiring hemodialysis or high-dose glucocorticoids such as prednisone of ≥ 100 mg/day (or other glucocorticoids with equivalent doses).
3. Cardiovascular disorders: history of acute myocardial infarction, or unstable angina, severe arrhythmia (multifocal frequent ventricular premature beats, ventricular tachycardia, ventricular fibrillation), etc. over the past six months; New York Heart Association (NYHA) Class III-IV (see Annex 6. NYHA for details).
4. Subjects with a known history of moderate or severe persistent asthma (assessed by the Asthma Severity Scale of the National Heart, Lung, and Blood Institute [NHLB]) within the past 5 years, or who currently have uncontrolled asthma (of any grade).
5. Asthma and specific dermatitis, etc. requiring glucocorticoid-dependent therapy (except topical glucocorticoids).
6. Infections, requiring treatment for acute or chronic infections, as follows:

   * Treatment with any inhibitory therapy currently for chronic infections (e.g., tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, zoster virus and atypical mycobacteriosis);
   * Hospitalization for an infection within 60 days prior to dosing;
   * Treatment with anti-infective drugs (antibacterials, antivirals, antifungals, or antiparasites) by parenteral administration (IV or IM) 60 days prior to dosing.
   * Subjects with mycobacterium tuberculosis, including those with a positive "T-cell spot test for tuberculosis infection (T-SPOT)" (latent tuberculosis infection: except those who have completed tuberculosis prophylaxis for 4 weeks before their first dose), or those with a positive imaging result.
7. Subjects with positive results from any of the following tests: hepatitis B surface antigen (HBs Ag), hepatitis B core antibody (HBc Ab), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus antibody (HIV Ab), or treponema pallidum antibody (TPPA). Patients who tested positive for hepatitis B core antibody (HBc Ab) but negative for HBV-DNA should be excluded.
8. Hematological system diseases or hematology abnormalities: subjects with previous or current hematological system diseases (including but not limited to: myelofibrosis, anemia aplastic aregenerative, leukemia, lymphoma, etc.), hematology with hemoglobin < 100 g/L, white blood cells < 3.0 × 109/L, granulocytes < 2.5 × 109/L, lymphocytes < 0.8 × 109/L, or platelets < 100 × 109/L.
9. Abnormal liver function: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or glutamyl transpeptidase (GGT) values > 2 times ULN; or total bilirubin or alkaline phosphatase (ALP) values > 1.5 times ULN.
10. Abnormal renal function: creatinine (Cr) or urea nitrogen (BUN) values > 1.5 times the upper limit of normal (ULN); pre-screening estimated glomerular filtration rate (eGFR) ≤ 60 mL/min. Calculate eGFR values using the MDRD formula: eGFR (mL/min × 1.73 m2) = 175 × blood creatinine ([Scr (mg/dL)])-1.154 × age-0.203 × sex (M = 1, F = 0.742).
11. Cancer: history of malignancy within the last 5 years.
12. Transplant: history of major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell or bone marrow transplant.
13. Female subjects with a positive serum pregnancy test or currently lactating.
14. History of major surgery (craniotomy, thoracotomy, or laparotomy) or presence of unhealed wounds, ulcers, or fractures within 4 weeks prior to the first dose of study treatment.
15. Targeted drug therapy: rituximab within 180 days before the first dose; any drug therapy targeting T-lymphocytes, B-lymphocytes, cytokines or receptors [e.g., belimumab, telitacicept, abatacept, etc.] within 90 days before the first dose; JAK inhibitors within 30 days before the first dose; other investigational drugs for less than 5 half-lives.
16. Subjects who have participated in any other clinical trials (including receiving investigational vaccines) or received treatment with invasive and investigational medical devices within 3 months before inclusion, or are being enrolled into an interventional and investigational study.
17. Stable doses of anticoagulant or antiplatelet drugs used before randomization that exceeded regular doses or was increased within 7 days before dosing.
18. Immunosuppressants:

    * Have received any of the following treatments within 90 days prior to screening: Intravenous immunoglobulin (IVIG);Use of high-dose glucocorticoids such as prednisone ≥ 100 mg/day;Plasma exchange, leukopheresis;Cyclophosphamide.
    * Use of immunomodulatory agents such as thymosin within 30 days prior to screening.
19. Vaccination within 30 days prior to the first dose of study treatment.
20. Use of traditional Chinese medicinal products or herbal preparations such as total glucosides of white paeony capsules, zhengqinfengtongning and colquhounia root tablets within 30 days prior to the first dose of study treatment.
21. Drug abusers determined by medication history inquiries, including morphine, ketamine, tetrahydrocannabinolate, methamphetamine, dimethyldioxymethamphetamine and cocaine.
22. Subjects who have consumed more than 14 units of alcohol/week (1 unit of alcohol = 360 mL of beer, 150 mL of wine, or 45 mL of liquor) within 3 months prior to screening, or who cannot abstain from alcohol during the trial, as determined by history inquiries.
23. Other conditions: including laboratory abnormalities, history of any other disease (e.g., recent history of septicemia), clinically significant unstable or uncontrolled acute or chronic conditions unrelated to SLE (e.g., acute pneumonia, pulmonary arterial hypertension, diabetic ketoacidosis, acute pancreatitis, etc.). In the opinion of the investigator, the above conditions may confound the study results or place the subject at an inappropriate risk. Thus, the subjects who experience the conditions above are not suitable for participation in this study.
24. Subjects who are unsuitable for participation in this clinical study for any other reasons as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Rate of Adverse Events | 43 days post last dose for single dose
  Evaluate the rate of adverse events
Rate of Adverse Events | 113 days post last dose for multi- dose
  Evaluate the rate of adverse events
Pharmacokinetic(PK) Parameters: Cmax | 43 days post last dose for single dose,
  Cmax
Pharmacokinetic(PK) Parameters: Cmax | 113 days post last dose for multi- dose
  Cmax
Pharmacokinetic(PK) Parameters: Tmax | 43 days post last dose for single dose,
  Tmax
Pharmacokinetic(PK) Parameters: Tmax | 113 days post last dose for multi- dose
  Tmax
Pharmacokinetic(PK) Parameters: AUC | 43 days post last dose for single dose,
  AUC0-tlast
Pharmacokinetic(PK) Parameters: AUC | 113 days post last dose for multi- dose
  AUC0-tlast

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hosptial Zhejiang University School of Medicine, Zhejiang, Hangzhou
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality